CLINICAL TRIAL: NCT01301924
Title: Phase III Clinical Trial for American Tegumentary Leishmaniasis: Comparison of Standard and Alternative Antimonial Dosage in Patients With American Cutaneous Leishmaniasis
Brief Title: Comparison of Standard and Alternative Antimonial Dosage in Patients With American Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, ASchubach, Senior Researcher, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StdvsaltCL
Record Dates: First submitted 2011-02-20; First posted 2011-02-23 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Leishmaniasis Cutaneous; Leishmania braziliensis; Meglumine Antimoniate; Treatment Effectiveness; Controlled Clinical Trials, Randomized
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate; Contraceptives, Oral

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose (Active Comparator): High dose: 20 days of 20 mg/kg/day meglumine antimoniate
  Interventions: Drug: Meglumine antimoniate
- Low dose (Experimental): Low dose: 30 days of 5 mg/kg/day meglumine antimoniate
  Interventions: Drug: Meglumine antimoniate

INTERVENTIONS:
Drug: Meglumine antimoniate — Meglumine antimoniate is stored and ministered under actual conditions employed by health services in Brazil. Each patient will be included in one of the treatment groups with meglumine antimoniate IM:
  High dose: 20 days of 20 mg/kg/day antimoniate meglumine. Low dose: 30 days of 5 mg/kg/day antimoniate meglumine.
  Other Names: High dose; Low dose

SUMMARY:
"Phase III Clinical Trial for American Tegumentary Leishmaniasis: Comparison of Standard and Alternative Antimonial Dosage in Patients With American Cutaneous Leishmaniasis " has begun in October 2008 at the Laboratory of Leishmaniasis Surveillance at Evandro Chagas Clinical Research Institute (IPEC), FIOCRUZ, aiming to compare efficacy and safety of the standard recommended schedule with an alternative dosage scheme of meglumine antimoniate in the treatment of American tegumentary leishmaniasis (ATL). It is a study with blind evaluation by the doctors and the responsible for statistical analysis. Patients diagnosed with ATL, eligible for the trial are randomly allocated into one of the schemes with meglumine antimoniate and monitored before, during and after it. There is no single regimen applicable to all forms of leishmaniasis around the world. Therapeutic regimens applied to treat people living in other geographic areas result in mixed outcomes. Ideally, the most appropriate regimens should be established for each endemic area, based on its efficacy, toxicity, difficulties of administration and cost. Given the problems and limitations of the use of pentavalent antimonials (Sb5+) at 20 mg Sb5+ / kg / day, less toxic alternative regimens, i.e. 5mg Sb5+/kg/day, deserve to be better evaluated. The treatment of ATL must heal skin lesions and prevent late mucosal lesion development. The indication of high doses of Sb5+ is based on the evidence that there could be induction of resistance with use of subdoses. However, clinical studies with extended follow-up in Rio de Janeiro have suggested that regular low doses (5mg Sb5+ / kg / day) may constitute an effective scheme, achieving cure rates similar to higher doses, with lower toxicity, ease of implementation and lower cost. Published studies on efficacy and safety of alternative dosage schemes with meglumine antimoniate failed to provide conclusive results so far, for various methodological biases. The need to compare the effectiveness and safety between the standard treatment scheme with meglumine antimoniate currently recommended in Brazil for the treatment of ATL and an alternative scheme with low doses of antimony is the motive for this study in Rio de Janeiro.

DETAILED DESCRIPTION:
1. Introduction. Pentavalent antimonials are first line drugs for the treatment of leishmaniasis. WHO and Brazilian Ministry of Health recommend treating patients with cutaneous leishmaniasis (CL) with doses of 20mg/kg/day, IM or IV, for three to four weeks. In the Reference Centre on Leishmaniasis - IPEC - FIOCRUZ, the dose of 5mg/kg/day IM has been effective and well tolerated in the treatment of CL. CL is treated for 30 days, with a lower incidence of adverse effects and lower treatment dropout rates. In all cases patients should be monitored with clinical examination, electrocardiogram (EKG), blood count, liver, renal and pancreatic function tests. Some side effects can be observed, although they not necessarily lead to discontinuation of treatment. EKG most frequent abnormalities are heart rhythm and disturbances of ventricular repolarization: flattening or inversion of T wave and adjusted QT space widening.
2. Background: Ideally, the most appropriate antimoniate therapeutic regimens should be established for each area, based on their efficacy and toxicity, without ignoring the difficulties of administration and cost. The treatment of CL must achieve healing of skin lesions and prevention of late mucosal involvement. The recognition, recommendation and acceptance of new regimens should be preceded by demonstration of their superiority to currently recommended treatments. We aim to compare the effectiveness and safety among treatment schemes with meglumine antimoniate currently recommended in Brazil for the treatment of CL and the alternative scheme with low dose of antimony.
3. Objectives. 3.1. General Objective. To compare the effectiveness and safety of 20 days of 20 mg/kg/day meglumine antimoniate with 30 days of 5 mg/kg/day meglumine antimoniate in the treatment of patients with CL.

   3.2. Specific Objectives. 3.2.1. To evaluate non-inferiority of low dose group as compared to the high dose antimonial therapy for CL.

   3.2.2. To compare the effectiveness immediately and up to two years after treatment, of the different groups of antimonial therapy for CL.

   3.2.3. To compare the frequency and severity of clinical, laboratory and EKG adverse events between different antimonial treatment groups.

   3.2.4. To compare the frequency and severity of adverse events between elderly and young people between the groups.

   3.2.5. To compare the frequencies of epithelialization achieved on days 20, 30 and 50 of treatment in each patient.

   3.2.6. To compare the time in days up to the epithelialization of the lesions according to location above and below the knees, controlling for concomitant vascular insufficiency.
4. Subjects and methods.

4. 1. Study design: Controlled clinical trial with standard treatment, randomized, single-blind, phase III.

4.2. Description of interventions: Meglumine antimoniate (Aventis, São Paulo, Brazil) is stored and ministered under actual conditions employed by the health services in Brazil. Each patient will be included in one of two treatment groups with meglumine antimoniate IM: a) 20 days of 20 mg/kg/day meglumine antimoniate, b) 30 days of 5 mg/kg/day meglumine antimoniate. There will be no cross-over between the groups for the purpose of this study. The data from those patients who require permanent discontinuation of a scheme will be assessed in the group that were randomized, ie, by modified intention to treat. Analysis will be performed by modified intention to treat and per protocol.

4.3. Sampling plan. 4.3.1 Sample size. The comparison of the effectiveness between the four schemes should reveal similar results for the following outcomes: a) frequency of good initial response; b) time (days) until the epithelialization of all lesions; c) time (days) to achieve the complete healing of all lesions; d) frequency of late response (two years of follow-up according to schedule); e) frequency of reactivation after treatment (up to 2 years of follow-up). With a significance level of 5% and 80% power to calculate the sample sizes to compare the groups; initially, a 60-total of patients will be required for non-inferiority analysis with a margin of 15%. For equivalence analysis, a 264-total of patients will be required.

4.4 Allocation strategy (randomization). Individuals eligible (see eligibility criteria) and who agree to participate (by signing an informed consent) will be randomly assigned to one of two treatment groups, according to order of arrival until the completion of the total groups.

4.5. Eligibility Criteria (see item: Eligibility Criteria). 4.6. Outcomes. 4.6.1 Effectiveness outcomes: Definition. a) Initial therapeutic response - presence or no of complete epithelialization of all lesions until day 110. b) Late therapeutic response - the presence or no of the following elements in the progression to healing: - disappearance of crusts until day 140; -disappearance of desquamation until day 230; - disappearance of infiltration until day 320; -disappearance of erythema until day 410; - no appearance of mucosal damage until day 770; - recurrence of any stage prior to that achieved and maintained in two observations with an interval of at least two weeks. 4.6.2 Safety outcomes (adverse events): definition, intensity and relationship to study drug. An adverse event (AE) is any effect, adverse or unexpected, evidenced by the investigator or reported by patients, beginning during the drug use or until 30 days after stopping it. The investigation of AE shall be made for both spontaneous recall and question by the physician according to a standardized form on days 10, 20, 30, 50, 60 and 80. The classification of the severity of adverse events (clinical, laboratory and electrocardiographic) will take place according to "AIDS Table for Grading Severity of Adult Adverse Experiences, 1992". The causal relationship to study drug (= AE) will be evaluated by the investigator and classified as follows: a) Definite (Highly Likely); b) Probable; c) Possible; d) Remote (Probably not); e) Definitely not.

4.7. Management of adverse effects. The AE will be noted in the appropriate form and shall contain: a description of the adverse effect, its intensity, relation with the investigated drug, start date, completion date, duration and conduct taken.

4.8. Masking. We chose to perform the measurements of outcomes of interest (effectiveness) and adverse events (clinical) by a physician who is not aware of what is the regimen used by the patient. It is intended to minimize measurement biases of the different outcomes according to treatment regimen to which each patient belongs. The results of laboratory tests are provided by the clinical pathology laboratory without information about the treatment group. The manager of database preserves the secrecy of this information by coding the groups for analysis for the epidemiologist(s).

4.9. Criteria for definitive discontinuation of study treatment: a) Interrupt driven by clinical, laboratory or EKG AE Grade 4; b) Interruption exceeding 10 days attributed to clinical, laboratory or EKG adverse event Grade <3; c) Spontaneous cessation of the use of prescribed medication beyond five consecutive doses, due to fault of the administration (noncompliance).

4.10. Criteria for study withdrawal: a) definitive interruption of treatment; b) Pregnancy; c) introduction of immunosuppressive drugs or potentially toxic; d) intercurrent disease, unrelated to study drug, but with demonstrations equivalent or superior to clinical grade 3 AE; e) poor initial or late therapeutic response; f) patient withdrawal to continue the study.

4.11. Procedures for confidentiality break. The randomization codes used for allocation of numbering and allocation of patients may be revealed in cases of necessity of the study.

4.12. Monitoring the study. The parameters (outcomes) of effectiveness and safety will be monitored according to the timetable for implementation. The principal investigator and coordinators will supervise the field work, controlling for quality deviation and this Protocol. Important items to be monitored: adhesion to the Protocol (follow-up losses will be minimized through active search), appropriate records of outcomes and adverse events; adequacy of stored products; quality of procedures for laboratory tests; minimization of missing data; periodic transmission of data for data entry. Written reports of field will be retained for consideration by the committees. Report of serious adverse events to the CEP/IPEC and decision to interrupt the test. External Committee: a committee of outside monitoring of the trial shall be constituted , consisting of three members, experts in the treatment of CL and execution of clinical trials. The committee will carry out audits of documentation and activities relevant to the clinical trial, controlling for possible protocol breaks.

4.13 Control of storage of medications. The ampoules required for complete treatment of the whole sample will be stored in the Pharmacy of IPEC. A trained team professional will include the patients, in day 1 consultation, following the randomization list.

4.14. Data Analysis Plan. Data analysis will be carried out following the principle of intention to treat. The data from those patients who require permanent discontinuation of a scheme will be analyzed according to the group for what they had been allocated initially, not being re-assigned to another group to resumption of treatment (no cross-over between the groups for the purpose of this study). We will describe the simple frequencies of categorical variables and measures of central tendency and dispersion of continuous quantitative variables for each antimony scheme. The proportion of dichotomous outcome of presence or absence of scarring in each group will be compared to the standard (chi-square) and through analysis of survival the time in days until reaching healing (log-rank statistic). The healing frequencies are compared by ratio test type chi-square, the median time to healing through comparison test of means (Student's t type) three or more (ANOVA) and survival analysis for outcomes that involve time in days, if necessary will be used nonparametric tests. To evaluate the efficacy and safety are also estimated the relative risk (RR) and the absolute risk reduction (ARR) and relative risk reduction (RRR). For paired comparison of proportions of healing on days 20, 30 and 50 will be employed the Mann-Whitney test 5. Ethical considerations. 6.1 Risks and benefits. The main potential benefit of this test is the possibility of subsidizing the use of lower doses of antimony, potentially less toxic and less costly. The risks consist of general adverse events, which will be thoroughly scrutinized and treated according to the schedule attached. This project was submitted to the Research Ethics Committee (CEP/IPEC) and CONEP. All patients sign an informed consent. This project follows the recommendations contained in the resolution 196/96 of the National Health Council.

5.2. Informed consent. In plain language and explaining the objectives, risks, benefits and identifying those responsible for research.

6. Expected Results. We hope that low dose is non inferior to the high dose antimonial treatment and that the different schemes are equivalent in effectiveness, and with diverse toxicities.

7. Financial support. This project is supported in part with funds approved by MCT/CNPq / MS-SCTIE-DECIT 25/2006.

ELIGIBILITY:
Eligibility Criteria.

Inclusion criteria:

1. Cutaneous leishmaniasis with parasitological diagnosis by one or more of the following methods: direct examination (scraping or imprint), histopathology, culture, immunohistochemistry, or PCR.
2. History of exposure in an endemic area of Rio de Janeiro
3. Absence of prior treatment with meglumine antimoniate

Exclusion criteria:

1. women who do not use contraceptives or do it inadequately
2. pregnant
3. under 13
4. prior treatment with meglumine antimoniate
5. use of immunosuppressive therapy (steroids, cancer chemotherapy) or medicines for tuberculosis or leprosy.
6. presence of changes in baseline clinical adverse effect level equivalent to> G3
7. presence of changes in baseline laboratory adverse effect level equivalent to> G2
8. presence of baseline electrocardiographic changes equivalent to an adverse effect level> G4 and / or baseline QTc> 0.46 ms (equivalent to AS level G1).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-10; Primary Completion 2016-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of meglumine antimoniate treatment | 6 years
  To compare the effectiveness of meglumine antimoniate at a dose of 5 mg or 20 mg Sb5+ / kg / day in the treatment of patients with cutaneous leishmaniasis.

SECONDARY OUTCOMES:
Safety of meglumine antimoniate treatment | 6 years
  To compare the safety of meglumine antimoniate at a dose of 5 mg or 20 mg Sb5+ / kg / day in the treatment of patients with cutaneous leishmaniasis.

CONTACTS AND LOCATIONS:
Overall Officials: Armando O. Schubach, MD, PhD, Study Director — IPEC/FIOCRUZ
Locations (1):
- Oswaldo Cruz Foundation - IPEC/FIOCRUZ, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antezana G, Zeballos R, Mendoza C, Lyevre P, Valda L, Cardenas F, Noriega I, Ugarte H, Dedet JP. Electrocardiographic alterations during treatment of mucocutaneous leishmaniasis with meglumine antimoniate and allopurinol. Trans R Soc Trop Med Hyg. 1992 Jan-Feb;86(1):31-3. doi: 10.1016/0035-9203(92)90427-e. PMID 1566297
- [Background] de Azeredo-Coutinho RB, Mendonca SC. An intermittent schedule is better than continuous regimen of antimonial therapy for cutaneous leishmaniasis in the municipality of Rio de Janeiro, Brazil. Rev Soc Bras Med Trop. 2002 Sep-Oct;35(5):477-81. doi: 10.1590/s0037-86822002000500009. PMID 12621667
- [Background] Chulay JD, Spencer HC, Mugambi M. Electrocardiographic changes during treatment of leishmaniasis with pentavalent antimony (sodium stibogluconate). Am J Trop Med Hyg. 1985 Jul;34(4):702-9. doi: 10.4269/ajtmh.1985.34.702. PMID 2992303
- [Background] Deps PD, Viana MC, Falqueto A, Dietze R. [Comparative assessment of the efficacy and toxicity of N-methyl-glucamine and BP88 sodium stibogluconate in the treatment of localized cutaneous leishmaniasis]. Rev Soc Bras Med Trop. 2000 Nov-Dec;33(6):535-43. doi: 10.1590/s0037-86822000000600004. Portuguese. PMID 11175583
- [Background] Hepburn NC, Nolan J, Fenn L, Herd RM, Neilson JM, Sutherland GR, Fox KA. Cardiac effects of sodium stibogluconate: myocardial, electrophysiological and biochemical studies. QJM. 1994 Aug;87(8):465-72. PMID 7922300
- [Background] Hepburn NC, Siddique I, Howie AF, Beckett GJ, Hayes PC. Hepatotoxicity of sodium stibogluconate therapy for American cutaneous leishmaniasis. Trans R Soc Trop Med Hyg. 1994 Jul-Aug;88(4):453-5. doi: 10.1016/0035-9203(94)90432-4. PMID 7570843
- [Background] Marzochi MC, Marzochi KB. Tegumentary and visceral leishmaniases in Brazil: emerging anthropozoonosis and possibilities for their control. Cad Saude Publica. 1994;10 Suppl 2:359-75. doi: 10.1590/s0102-311x1994000800014. Epub 2004 Mar 19. PMID 15042226
- [Background] McBride MO, Linney M, Davidson RN, Weber JN. Pancreatic necrosis following treatment of leishmaniasis with sodium stibogluconate. Clin Infect Dis. 1995 Sep;21(3):710. doi: 10.1093/clinids/21.3.710. No abstract available. PMID 8527590
- [Background] Oliveira Neto MP, Schubach A, Araujo ML, Pirmez C. High and low doses of antimony (Sbv) in American cutaneous leishmaniasis. A five years follow-up study of 15 patients. Mem Inst Oswaldo Cruz. 1996 Mar-Apr;91(2):207-9. doi: 10.1590/s0074-02761996000200016. PMID 8736092
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, da Costa SC, Pirmez C. Intralesional therapy of American cutaneous leishmaniasis with pentavalent antimony in Rio de Janeiro, Brazil--an area of Leishmania (V.) braziliensis transmission. Int J Dermatol. 1997 Jun;36(6):463-8. doi: 10.1046/j.1365-4362.1997.00188.x. PMID 9248897
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, Goncalves-Costa SC, Pirmez C. A low-dose antimony treatment in 159 patients with American cutaneous leishmaniasis: extensive follow-up studies (up to 10 years). Am J Trop Med Hyg. 1997 Dec;57(6):651-5. doi: 10.4269/ajtmh.1997.57.651. PMID 9430521
- [Background] Oliveira-Neto MP, Schubach A, Mattos M, Goncalves-Costa SC, Pirmez C. Treatment of American cutaneous leishmaniasis: a comparison between low dosage (5 mg/kg/day) and high dosage (20 mg/kg/day) antimony regimens. Pathol Biol (Paris). 1997 Jun;45(6):496-9. PMID 9309267
- [Background] Ribeiro AL, Drummond JB, Volpini AC, Andrade AC, Passos VM. Electrocardiographic changes during low-dose, short-term therapy of cutaneous leishmaniasis with the pentavalent antimonial meglumine. Braz J Med Biol Res. 1999 Mar;32(3):297-301. doi: 10.1590/s0100-879x1999000300008. PMID 10347787
- [Background] Rodrigues ML, Costa RS, Souza CS, Foss NT, Roselino AM. Nephrotoxicity attributed to meglumine antimoniate (Glucantime) in the treatment of generalized cutaneous leishmaniasis. Rev Inst Med Trop Sao Paulo. 1999 Jan-Feb;41(1):33-7. doi: 10.1590/s0036-46651999000100007. PMID 10436668
- [Background] Sampaio RN, de Paula CD, Sampaio JH, Furtado Rde S, Leal PP, Rosa TT, Rodrigues ME, Veiga JP. [The evaluation of the tolerance and nephrotoxicity of pentavalent antimony administered in a dose of 40 mg Sb V/kg/day, 12/12 hr, for 30 days in the mucocutaneous form of leishmaniasis]. Rev Soc Bras Med Trop. 1997 Nov-Dec;30(6):457-63. doi: 10.1590/s0037-86821997000600003. Portuguese. PMID 9463192
- [Background] Schubach Ade O, Marzochi KB, Moreira JS, Schubach TM, Araujo ML, Vale AC, Passos SR, Marzochi MC. Retrospective study of 151 patients with cutaneous leishmaniasis treated with meglumine antimoniate. Rev Soc Bras Med Trop. 2005 May-Jun;38(3):213-7. doi: 10.1590/s0037-86822005000300001. Epub 2005 May 4. PMID 15895170
- [Background] Sharquie KE. A new intralesional therapy of cutaneous leishmaniasis with hypertonic sodium chloride solution. J Dermatol. 1995 Oct;22(10):732-7. doi: 10.1111/j.1346-8138.1995.tb03911.x. PMID 8586751
- [Background] Veiga JP, Wolff ER, Sampaio RN, Marsden PD. Renal tubular dysfunction in patients with mucocutaneous leishmaniasis treated with pentavalent antimonials. Lancet. 1983 Sep 3;2(8349):569. doi: 10.1016/s0140-6736(83)90595-0. No abstract available. PMID 6136717
- [Derived] Saheki MN, Lyra MR, Bedoya-Pacheco SJ, Antonio LF, Pimentel MIF, Salgueiro MM, Vasconcellos ECFE, Passos SRL, Santos GPLD, Ribeiro MN, Fagundes A, Madeira MF, Mouta-Confort E, Marzochi MCA, Valete-Rosalino CM, Schubach AO. Low versus high dose of antimony for American cutaneous leishmaniasis: A randomized controlled blind non-inferiority trial in Rio de Janeiro, Brazil. PLoS One. 2017 May 30;12(5):e0178592. doi: 10.1371/journal.pone.0178592. eCollection 2017. PMID 28558061
- See also: Oswaldo Cruz Foundation is responsible for a range of activities which include research development; production of vaccines, drugs, reagents, etc; quality control of products and services; education and the implementation of social programs. — http://www.fiocruz.br
- See also: Evandro Chagas Clinical Research Institute (IPEC), FIOCRUZ — http://www.ipec.fiocruz.br